CLINICAL TRIAL: NCT03848390
Title: Effect of Modified Time-restricted Feeding in Preventing Progression of Non-Alcoholic Fatty Liver Disease (NAFLD).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Essam M. Imseis, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-1022
Record Dates: First submitted 2019-02-08; First posted 2019-02-20 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Time-restricted Feeding (Experimental)
  Interventions: Behavioral: Modified Time-restricted Feeding; Behavioral: Physical activity; Behavioral: Restricted consumption of sweetened beverages
- Conventional diet (Active Comparator)
  Interventions: Behavioral: Conventional diet; Behavioral: Physical activity; Behavioral: Restricted consumption of sweetened beverages

INTERVENTIONS:
Behavioral: Conventional diet — The conventional diet arm will be asked to consume a hypocaloric diet, and they will be allowed to eat at any time of the day with no time restriction.
  Arms: Conventional diet
Behavioral: Modified Time-restricted Feeding — The modified time-restricted feeding arm will be asked to consume any food but will be asked to consume this food for only a 9 hour daytime period.
  Arms: Modified Time-restricted Feeding
Behavioral: Physical activity — At least 30 minutes of physical activity per day 5 times per week.
Behavioral: Restricted consumption of sweetened beverages — Restricted consumption of juice, soda, and other sweetened beverages.

SUMMARY:
The purpose of the study is to examine the effects of modified time-restricted feeding and conventional dietary approaches in motivated obese fatty liver patients on biochemical markers, imaging studies, and anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Motivated obese fatty liver patients aged 8 -18yrs with ALT >80

Exclusion Criteria:

* Patients with metabolic disorders,
* On certain medications (i.e., amiodarone, corticosteroids, methotrexate, select antipsychotics /antidepressants, HAART, valproic acid),
* Kwashiorkor
* Alcohol abuse,
* Rapid surgical weight loss,
* History of parenteral nutrition and
* Hepatitis C.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Alanine Amino Transferase (ALT) levels | Baseline, 3 months

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) Z-score | Baseline, 3 months
Change in hepatic steatosis on Magnetic Resonance Elastography of the Liver | Baseline, 3 months
Change in fibrosis on Magnetic Resonance Elastography of the Liver | Baseline, 3 months
Change in diastolic blood pressure | Baseline, 3 months
Change in systolic blood pressure | Baseline, 3 months
Change in LDL | Baseline, 3 months
Change in HDL | Baseline, 3 months
Change in TRIGLYCERIDE | Baseline, 3 months
Change in TOTAL CHOLESTEROL | Baseline, 3 months
Hemoglobin A1C | Baseline; 3 months
Fasting serum insulin | Baseline; 3 months
Fasting serum glucose | Baseline; 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Essam M Imseis, MD, Principal Investigator — The University of Texas Health Sciences Center in Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No